CLINICAL TRIAL: NCT07013279
Title: A Double-blind, Randomized, Active-controlled, Multi-center, Phase III Study to Evaluate the Efficacy and Safety of DWP712 Inj. in Subjects With Moderate to Severe Glabellar Lines
Brief Title: Evaluate the Efficacy and Safety of DWP712 With Moderate to Severe Glabellar Lines
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW_DWP712301
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Glabellar Lines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DWP712 inj. (Experimental): The investigational product will be administered by a single intramuscular injection, and 4 U/0.1 mL of the IP will be injected into a total of 5 sites, totaling 20 U/0.5 mL.
  Interventions: Biological: DWP712 inj.
- Botox® 100 Units (Active Comparator): The investigational product will be administered by a single intramuscular injection, and 4 U/0.1 mL of the IP will be injected into a total of 5 sites, totaling 20 U/0.5 mL.
  Interventions: Biological: Botox® 100 Units

INTERVENTIONS:
Biological: DWP712 inj. — Clostridium botulinum Toxin
  Arms: DWP712 inj.
Biological: Botox® 100 Units — Clostridium botulinum Toxin
  Arms: Botox® 100 Units

SUMMARY:
To evaluate the efficacy and safety of DWP712 Inj. in Subjects with Moderate to Severe Glabellar Lines

ELIGIBILITY:
Inclusion Criteria:

- Subjects with a facial wrinkle scale (FWS) score of ≥2 (moderate) for glabellar lines at maximum frown in the investigator's on-site assessment at screening

Exclusion Criteria:

- Subjects with glabellar lines that cannot sufficiently be improved by physical attempts, e.g., glabellar lines not flattened by hand, in the judgment of the investigator

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects with glabellar line improvement* rate at maximum frown based on the investigator's on-site assessment at 4 weeks after IP administration | At 4 weeks after IP administration
  Improvement means FWS grade of "0" or "1" with a ≥2-point improvement from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Chung-Ang University Hosptial, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No